CLINICAL TRIAL: NCT01572805
Title: Evaluation of Melatonin's Effect on Pain and Blood Loss After Cesarean Section
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, marzieh beigom khezri, Assistant professor, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACTRN12612000117819
Record Dates: First submitted 2012-04-03; First posted 2012-04-06 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Post Partum Haemorrhage in Patients Undergoing Cesarean Section
Keywords: Post partum haemorrhage; Cesarean; Pain
MeSH Terms: conditions — Postpartum Hemorrhage; Pain | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- melatonin 3mg (Active Comparator)
  Interventions: Drug: melatonin 3mg
- melatonin 6mg (Active Comparator)
  Interventions: Drug: melatonin 6mg
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: melatonin 3mg — To receive sublingual 3 mg melatonin before spinal of anesthesia .
  Arms: melatonin 3mg
Drug: melatonin 6mg — To receive sublingual 6 mg melatonin before spinal of anesthesia .
  Arms: melatonin 6mg
Drug: placebo — To receive sublingual placebo tablet before spinal of anesthesia .
  Arms: placebo

SUMMARY:
The purpose of this study is to assess the effect of melatonin on pain and amount of blood loss after cesarean delivery one hundred twenty women with singleton term pregnancy undergoing elective or emergency lower segment cesarean section under spinal anesthesia were included in this study. The patients were randomly allocated to one of three groups of 40 each to receive sublingual 3 mg melatonin or 6 mg melatonin or placebo before spinal of anesthesia . In all patients 20 IU syntocinon which dissolved in 0.5liter of lactated Ringer's solution) at the rate of 500 ml over a 15 minutes period, immediately after delivery of the neonate was infused . Time to first requirement of analgesic supplement, Hemodynamic variables,will be recorded.Patients were instructed preoperatively in the use of the verbal rating scale (VRS) from 0 to 10 (0no pain, 10maximum imaginable pain) for pain assessment. If the VRS exceeded four and the patient requested a supplement analgesic, diclofenac Na supp 100 mg was to be given for post-operative pain relief as needed . For breakthrough pain(VRS >4) if time of administration of diclofenac Na less than 8h,Pethidine 25 mg IV was given. For determination of blood loss ,change in hemoglobin levels, need for additional oxytocics and ,the volume of blood in the suction bottle was measured, blood soaked sponges. Hemoglobin values were determined both before surgery and 12 h following surgery

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at term (37-40 wks) gestation scheduled for either elective or emergency lower segment cesarean section

Exclusion Criteria:

* women with any risk factor associated with an increased risk of postpartum hemorrhage were excluded i.e. multiple gestation, antepartum hemorrhage,poly-hydramnios, two or more previous cesarean sections and/or a history of previous rupture uterus
* current or previous history of significant disease including heart disease, liver, renal disorders ,anemia (Hb8 g%)or known coagulopathy

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Time to first requirement of analgesic supplement | Time to first requirement of analgesic supplement within 24 hours after intratechal injection
amount of blood loss after cesarean delivery | during surgery

SECONDARY OUTCOMES:
hemodynamic variables | 5min before the intrathecal injection,and at 2, 4, 6, 10, 15,20 min after the injection

CONTACTS AND LOCATIONS:
Locations (1):
- Qazvin Medical Science University, Qazvin, Qazvin Province, Iran

REFERENCES:
- [Derived] Khezri MB, Reihany MD, Dabbaghi Ghaleh T, Mohammadi N. Effect of Melatonin on Blood Loss After Cesarean Section: A Prospective Randomized Double-Blind Trial. J Obstet Gynaecol India. 2019 Oct;69(5):436-443. doi: 10.1007/s13224-019-01205-7. Epub 2019 Apr 24. PMID 31598047